CLINICAL TRIAL: NCT07289321
Title: Effect of Tramadol or Magnesium in Local Anesthetic Solution on Ultrasound-guided Bilateral TAP Block During Robotic Radical Prostatectomy on Acute Perioperative Pain and Chronic Postoperative Pain.
Brief Title: Tramadol / Magnesium in Ropivacaine Solution in UG-bilateral TAP Block and Analgesia in Robotic Radical Prostatectomy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Eftychios Stavroulakis, Anesthesiologist, MD, DESA, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 715/28-11-2025
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Perioperative Pain in Robotic Prostatectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Team A - ropivacaine solution for bilateral TAP block (Other): 30 Patients named team A will be administered an ultrasound-guided bilateral TAP block under aseptic conditions. The injected solution will contain 57 ml ropivacaine 0,375% plus 3 ml normal saline 0.9% and the needle used will be 20G 100mm. Both the total volume of the solution and the total amount of ropivacaine administered to all patients will be practically the same. Epinephrine will also be added to the local anesthetic solution so that the concentration will be 1:200,000. First of all, all the patients will receive general anesthesia and they will not differ in any way in terms of the doses (mg/kg) of medication they will receive for induction of anesthesia (according to their weight).
  Interventions: Other: Ultrasound - guided bilateral transversus abdominis plane block (TAP) in patients undergoing robotic-assisted radical prostatectomy.
- Team B - ropivacaine plus tramadol solution for bilateral TAP block (Active Comparator): 30 patients will receive a bilateral TAP block before robotic prostatectomy. The solution administered will be consisting of 57ml ropivacaine 0,375% plus 3 ml of tramadol (total dose 100mg) plus epinephrine 1:200.000 All the other conditions will be exactly the same.
  Interventions: Other: Ultrasound - guided bilateral transversus abdominis plane block (TAP) in patients undergoing robotic-assisted radical prostatectomy.
- Team C - ropivacaine plus magnesium solution for bilateral TAP block (Active Comparator): 30 patients will receive TAP block and the injected solution will be consisting 57ml ropivacaine 0,375% plus 3ml containing 300mg magnesium plus epinephrine 1:200.000
  Interventions: Other: Ultrasound - guided bilateral transversus abdominis plane block (TAP) in patients undergoing robotic-assisted radical prostatectomy.

INTERVENTIONS:
Other: Ultrasound - guided bilateral transversus abdominis plane block (TAP) in patients undergoing robotic-assisted radical prostatectomy. — 90 patients will be enrolled and divided in three different groups receiving U/G bilateral TAP block under aseptic conditions after induction of anesthesia and before the beginning of the surgery. The three groups of 30 patients each will differ in terms of the composition of the solution administered to them, in order to investigate any effect of 100mg tramadol or 300mg magnesium on the duration and the quality of the field block provided by ropivacaine injection. Both the total volume of the solution and the total amount of ropivacaine administered to all patients will be practically the same. Epinephrine will also be added to the local anesthetic solution so that the concentration will be 1:200,000. First of all, all the patients will receive general anesthesia and they will not differ in any way in terms of the doses (mg/kg) of medication they will receive for induction of anesthesia (according to their weight).

SUMMARY:
Tramadol and magnesium have already been researched in recent decades for their different roles in pain control. This clinical study will compare and re-evaluate their effect on the duration and quality of regional anesthesia technique. Participants will be men 40 to 80 years old with prostate cancer who are about to have robot-assisted radical prostatectomy. Initially, all males will be anaesthetised and then they will be randomly divided into three groups to undergo bilateral transverse abdominal plane (TAP) block under aseptic conditions. This involves insertion of a needle into the plane between internal oblique and transverse abdominal muscles under ultrasound guidance in order to inject the local anesthetic solution to relieve pain, as the responsible nerves run through the muscles of the abdominal wall. Specifically, 30 patients will receive only local anesthetic (ropivacaine), 30 will receive ropivacaine plus tramadol, and 30 will receive ropivacaine plus magnesium. Both the researchers and the participants will be unaware of (blind trial) the composition of the solution they will receive (double-blind randomized controlled trial). There will be no other differences in the other medications they will receive until the end of the surgery. Information will be collected in terms of the consumption of analgesic drugs both perioperatively and postoperatively (the first 24 hours of hospitalization), while the intensity of postoperative pain will also be assessed on a simple scale from 1 to 10 (Numerical Rating Scale - NRS). In addition, researchers will contact participants after 3 and 6 months to request an overall assessment of pain. The study will be conducted at the Aretaieio University Hospital in Athens, under the supervision of Anesthesiology Professors and will help us better understand the role of analgesic drugs already used in robotic surgery, which in the long term will contribute to the further development of even more effective protocols for the treatment of acute and chronic surgical pain. In general, the study is expected to last 3 years, which is the time required for patient enrollment, assessment of postoperative pain at 3 and 6 months, collection and analysis of all data. There are no additional risks or costs beyond those normally associated with radical prostatectomies, as nerve blocks (including TAP block) have already been adopted as analgesic methods at Aretaieio Hospital.

ELIGIBILITY:
Inclusion Criteria:

* males
* age 40-80 years
* physical status I-III according to the American Society of Anesthesiologists (ASA physical status)
* undergoing robotic-assisted radical prostatectomy using Da Vinci Xi.

Exclusion Criteria:

* Patients allergic to ropivacaine, tramadol, magnesium, or other drugs used in the study
* with coagulation disorders due to disease or medication,
* inflammation at the site of the block,
* addiction to alcohol
* history of opioid tolerance
* patients unable to complete the pain assessment scale
* patients unable or unwilling to provide written consent to participate in the study.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2028-12-10 (Estimated); Study Completion 2028-12-10 (Estimated)

PRIMARY OUTCOMES:
Perioperative fentanyl intravenous administration to patients. | According to Nociception level (NOL) algometry during general anesthesia for the robotically assisted radical prostatectomy.
  Minimal dose 2 μg/kg.
Τotal consumption of intravenous tramadol. | During the postoperative hospitalization of patients in the clinic in the first 24 hours after the end of the operation and the time of the first administration of tramadol.

SECONDARY OUTCOMES:
Intensity of acute postoperative pain according to numeric rating scale (NRS) and patient's overall satisfaction at 24 hours after surgery. | The assessment of the intensity of acute postoperative pain will be performed in the post-anesthesia care unit at 5, 15, 30, and 60 minutes and then in the ward at 2, 4, 8, and 24 hours after surgery.
Postoperative nausea and vomiting (PONV). | During the 24 hours postoperative hospitalisation of patients.

OTHER OUTCOMES:
Episodes of bradycardia or hypotension. | Perioperatively after TAP block administration.

CONTACTS AND LOCATIONS:
Overall Officials: Aikaterini Melemeni, Anaesthetist, Study Director — Aretaieion University Hospital
Locations (1):
- Aretaieion University Hospital of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided